CLINICAL TRIAL: NCT01692171
Title: Pharmacodynamics Study of Enoxalow, Produced by Blau Farmacêutica S/A, Compared to Clexane, Produced by Sanofi-Aventis Farmacêutica Ltda, in Healthy Subjects After Intravenous Administration.
Brief Title: Pharmacodynamics Study of Enoxalow Compared to Clexane in Healthy Subjects After Intravenous Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: Blau Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ENOBLA0612IV-I; Versão 01 datada de 20.06.2012 (Other: LAL Clinica)
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Healthy
Keywords: Subjects
MeSH Terms: interventions — Heparin, Low-Molecular-Weight; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teste (Experimental): Enoxalow (Heparin, Low-Molecular-Weight) - Blau Farmacêutica S/A.
  Interventions: Drug: Heparin, Low-Molecular-Weight
- Comparador (Active Comparator): Clexane (Heparin, Low-Molecular-Weight)- Sanofi-Aventis
  Interventions: Drug: Heparin, Low-Molecular-Weight

INTERVENTIONS:
Drug: Heparin, Low-Molecular-Weight — single intravenous administration of 3mg/Kg of the test drug and the comparator drug, according to randomization, in a crossover design, each administration separated by 6 days of washout.
  Other Names: Clexane; Enoxalow

SUMMARY:
The hypothesis of this trial is that the test drug (Enoxalow® - T) pharmacodynamics parameters are similar to the comparator drug (Clexane® - C) in healthy subjects following administration of single intravenous dose. The objective of this randomized, crossover, clinical trial is to evaluate the pharmacodynamic profile of the test drug Enoxalow® - T produced by Blau Farmacêutica, compared to the comparator drug Clexane®, produced by Sanofi-Aventis, by determining pharmacodynamic activities (including anti FXa and anti-FIIa), as surrogate markers for their circulating concentrations of the drug.

DETAILED DESCRIPTION:
In addition other pharmacodynamic tests such as Tissue Factor Pathway Inhibitor (TFPI) activity, as well as the ratio of anti-FXa and anti-FIIa activity will be compared as secundary obectives.

ELIGIBILITY:
Inclusion Criteria:

* Agree to all the purposes of the study by signing and dating the Informed Consent;
* Male, aged between 18 and 55 years, clinically healthy;
* BMI between 18.5 and 30;

Exclusion Criteria:

* Participation in clinical trials in the 12 months preceding the trial;
* Presence of pulmonary, cardiovascular, neurological, endocrine, gastrointestinal, genitourinary or other systems diseases;
* Acute disease in the period of 07 days before the beginning of the practical phase (administration of the drug) of the study;
* Chronic administration of medications for hypertension, diabetes or any other disease that requires continuous use of any drug;
* Hemoglobin <13 g/dL;
* Continuous use of oral anticoagulants, platelet inhibitors or anti-inflammatory drugs;
* Use of medications that interact with enoxaparin;
* History of gastrointestinal bleeding, deep vein thrombosis or pulmonary embolism that may interfere with the clinical outcome of the study;
* History of coagulopathy and bleeding diathesis;
* Presence of changes in physical examination suggestive of coagulation disorders (bruising, petechiae, or bruising);
* Body weight < 45 kg or > 100 kg;
* Absolute platelet count below 100 x 109 / L;
* History of chronic bleeding;
* History of acute haemorrhage in the past 30 days;
* History of sensitivity to mammalian-derived biological products, albumin or any component of the formulation;
* History of allergy or Steven Johnson disease;
* Current or previous history (under 12 months) use of illicit drugs and tobacco;
* History of alcohol abuse, current or previous (within 12 months);
* At the discretion of the Principal Investigator of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2013-10-31 (Actual)

PRIMARY OUTCOMES:
Assess the pharmacodynamic profile of the drug test in comparison to the comparator through the measurement of the activity of the Anti-FXa and anti-FIIa markers | The day after admission
  Post drug administration blood samples were collected at following times - 0; 0:10; 0:20; 0:30; 00:40 12:50; 1; 1:30; two; 2:30; 3; 3:30; 4; 5; 6; 8; 10; 12; 16:24 (± 30) hours after.

SECONDARY OUTCOMES:
Assess the pharmacodynamic profile of the drug test in comparison to the comparator through the measurement of the activity of the TFPI marker and ratio of Anti-FXa and anti-FIIa. | The day after admission
  Post drug administration blood samples were collected at following times - 0; 0:10; 0:20; 0:30; 00:40 12:50; 1; 1:30; two; 2:30; 3; 3:30; 4; 5; 6; 8; 10; 12; 16:24 (± 30) hours after.

CONTACTS AND LOCATIONS:
Overall Officials: Márcia Guidone, manager, Study Director — Blau Farmaceutica S.A.
Locations (1):
- LAL Clinica, Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bara L, Billaud E, Gramond G, Kher A, Samama M. Comparative pharmacokinetics of a low molecular weight heparin (PK 10 169) and unfractionated heparin after intravenous and subcutaneous administration. Thromb Res. 1985 Sep 1;39(5):631-6. doi: 10.1016/0049-3848(85)90244-0. No abstract available. PMID 4082105
- [Background] Bruno R, Baille P, Retout S, Vivier N, Veyrat-Follet C, Sanderink GJ, Becker R, Antman EM. Population pharmacokinetics and pharmacodynamics of enoxaparin in unstable angina and non-ST-segment elevation myocardial infarction. Br J Clin Pharmacol. 2003 Oct;56(4):407-14. doi: 10.1046/j.1365-2125.2003.01904.x. PMID 12968985
- [Background] EMA 2009. European Medicines Agency.Guideline on non-clinical and clinical development of similar biological medical products containing low-molecular-weightheparins:EMEA/CHMP/BMWP/118264/2007.
- [Background] FDA 2011. Food and Drug Administration. Draft Guidance on Enoxaparin Sodium.
- [Background] Gerotziafas GT, Petropoulou AD, Verdy E, Samama MM, Elalamy I. Effect of the anti-factor Xa and anti-factor IIa activities of low-molecular-weight heparins upon the phases of thrombin generation. J Thromb Haemost. 2007 May;5(5):955-62. doi: 10.1111/j.1538-7836.2007.02477.x. PMID 17461929
- [Background] Hirsh J, Warkentin TE, Shaughnessy SG, Anand SS, Halperin JL, Raschke R, Granger C, Ohman EM, Dalen JE. Heparin and low-molecular-weight heparin: mechanisms of action, pharmacokinetics, dosing, monitoring, efficacy, and safety. Chest. 2001 Jan;119(1 Suppl):64S-94S. doi: 10.1378/chest.119.1_suppl.64s. No abstract available. PMID 11157643
- [Background] Kuczka K, Harder S, Picard-Willems B, Warnke A, Donath F, Bianchini P, Parma B, Blume H. Biomarkers and coagulation tests for assessing the biosimilarity of a generic low-molecular-weight heparin: results of a study in healthy subjects with enoxaparin. J Clin Pharmacol. 2008 Oct;48(10):1189-96. doi: 10.1177/0091270008322911. Epub 2008 Aug 20. PMID 18716314
- [Background] Mousa SA, Bozarth J, Barrett JS. Pharmacodynamic properties of the low molecular weight heparin, tinzaparin: effect of molecular weight distribution on plasma tissue factor pathway inhibitor in healthy human subjects. J Clin Pharmacol. 2003 Jul;43(7):727-34. PMID 12856386
- [Background] Wannmacher L. Heparinas de baixo peso molecular: evidências que fundamentam indicações. Uso Racional de Medicamentos: Temas Selecionados 2007:4:1-6.